CLINICAL TRIAL: NCT07362953
Title: Paraclinical Assessment of Cardiometabolic Risk Based on Novel Biochemical İndices in Type 2 Diabetes
Brief Title: Paraclinical Cardiometabolic Risk Assessment in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Elif Azize Özşahin Delibaş, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-042
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Type 2 Diabetes; Metabolic-inflammatory indices
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus Group: Participants diagnosed with Type 2 Diabetes Mellitus who were included for baseline data collection.

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by impaired insulin action and increased cardiometabolic risk. Visceral adiposity, insulin resistance, systemic inflammation, and dyslipidemia play key roles in the development of cardiovascular disease in individuals with T2DM. In this context, simple, rapid, and cost-effective biomarkers are increasingly important for risk assessment. The triglyceride-glucose (TyG) index is a practical indicator of insulin resistance, while the Atherogenic Plasma Index (API) reflects cardiovascular risk related to dyslipidemia. The Systemic Immune Inflammation Index (SII), derived from routine blood counts, serves as a marker of systemic inflammation. This study aims to evaluate the predictive value of TyG, API, and SII in assessing insulin resistance, cardiometabolic risk, and inflammation in patients with T2DM, thereby supporting early diagnosis and improved clinical management.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic metabolic disorder characterized by the inability to adequately utilize essential nutrients, including carbohydrates, fats, and proteins, as a result of insulin deficiency and/or impaired insulin action. In individuals with type 2 diabetes mellitus (T2DM), comprehensive assessment of cardiovascular disease risk factors and visceral adiposity is of critical importance. Excess visceral fat is closely associated with increased insulin resistance and an elevated risk of cardiovascular disease, reflecting the well-established relationship between cardiometabolic disorders and adiposity. Moreover, excessive body fat accumulation contributes to a chronic low-grade systemic inflammatory state, which plays a central role in the pathogenesis of metabolic syndrome. When metabolic syndrome coexists with dyslipidemia, the risk of cardiovascular disease is further amplified.

In this context, the availability of biomarkers that are easy to apply, rapidly measurable, and cost-effective is of considerable clinical relevance. The triglyceride-glucose (TyG) index has emerged as a practical and reliable parameter for the assessment of insulin resistance. This index is calculated using fasting plasma triglyceride and glucose concentrations, which are routinely measured and widely accessible laboratory parameters. The TyG index provides valuable insight into metabolic disturbances related to insulin resistance and its potential association with cardiovascular disease. The Systemic Immune Inflammation Index (SII) is another emerging biomarker derived from peripheral blood cell counts, calculated using lymphocyte (L), platelet (P), and neutrophil (N) values, and reflects the balance between inflammatory and immune responses. In addition, the Atherogenic Plasma Index (API) serves as an indicator of atherogenic dyslipidemia and may offer information regarding the severity of insulin resistance associated with impaired glucose metabolism, as well as its relationship with cardiovascular risk.

The aim of this study is to evaluate the TyG index as a predictor of insulin resistance, the API as a marker of cardiovascular risk, and the SII as a significant indicator of systemic inflammation in patients diagnosed with T2DM. These novel biochemical indices may facilitate early risk stratification, improve treatment planning, and ultimately contribute to more effective clinical management of individuals with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of T2DM
* Having a diagnosis of prediabetes
* Being between 18 and 65 years of age.

Exclusion Criteria:

* Having any other chronic disease accompanying T2DM/prediabetes
* Receiving hormone therapy
* Using lipid-lowering agents
* Being pregnant/breastfeeding
* Having an acute infection
* Having any malignant/inflammatory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of type 2 diabetes mellitus or prediabetes attending the Department of Internal Medicine at Tokat Gaziosmanpaşa University Hospital during the study period will constitute the study population. Enrollment will be limited to individuals who meet the eligibility criteria and provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 2188 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Outcome Measure Title: Triglyceride-glucose index (TyG indice) | Description: Calculated using fasting glucose and triglyceride levels. Time Frame: At baseline Unit of Measure: Index value Calculated from hematological and biochemical results obtained by trained staff.
  TyG index: ln [fasting triglycerides (mg/dL) × fasting glucose (mg/dL)] / 2
Outcome Measure Title: Atherogenic Plasma Index (API) | Description: Calculated using HDL-cholesterol and triglycerides levels. Time Frame: At baseline Unit of Measure: Index value Calculated from hematological and biochemical results obtained by trained staff.
  API: log [triglycerides (mg/dL) / HDL-cholesterol (mg/dL)]
Outcome Measure Title: Systemic Immuno-Inflammation Index (SII) | Description: Calculated using platelet count, neutrophil count, lymphocyte count. Time Frame: At baseline Unit of Measure: Index value Calculated from hematological and biochemical results obtained by trained staff.
  SII = Platelet count x Neutrophil count / Lymphocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Delibaş, Principal Investigator — Tokat Gaziosmanpaşa Üniversitesi
Locations (1):
- Tokat Gaziosmanpaşa University Health Research and Application Hospital, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No